CLINICAL TRIAL: NCT06360822
Title: Increasing Equity in Lung Cancer Screening
Acronym: LUCARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eskenazi Health (Other)
Responsible Party: Principal Investigator, Nicholas Pettit, Principal Investigator, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19317
Record Dates: First submitted 2024-03-25; First posted 2024-04-11 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients will be shown a modified version of LungTalk.
  Interventions: Behavioral: ED-LCS
- Usual Care (No Intervention): Patients will receive usual care.

INTERVENTIONS:
Behavioral: ED-LCS — This is a lung cancer educational intervention for patients in the emergency department.
  Arms: Intervention

SUMMARY:
The overall objective of this mixed methods study is to: 1) Refine the Emergency Department Lung Cancer Screening (ED-LCS) intervention using qualitative interviews among key stakeholders; 2) pilot test the ED-LCS intervention evaluating the intervention efficacy, acceptability, and feasibility; and 3) provide an in-depth description of stakeholders' experiences with the ED-LCS intervention for future refinement.

ELIGIBILITY:
Inclusion Criteria:

* • Eligible for LCS (50-80 years old, smoked in past 15 years, and smoked at least 20 pack years)

Exclusion Criteria:

* • Non-English/Spanish speaking

  * Decompensated psychiatric illness (suicidal, homicidal, psychosis). Will confirm with attending physicians at time of enrollment
  * Intoxicated with alcohol or drugs
  * Cannot provide reliable follow up contact information (cell phone)
  * Presenting to the ED with a life-threatening condition
  * Have received chest CT scan in past 12 months
  * Already enrolled in LCS
  * Hospice enrolled

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of patients receive Lung Cancer Screening | 6-12 months

SECONDARY OUTCOMES:
Patients ratings of intervention | At delivery
  This is a subjective rating provided by patients of the intervention received

CONTACTS AND LOCATIONS:
Locations (1):
- Eskenazi Health, Indianapolis, Indiana, United States